CLINICAL TRIAL: NCT03686137
Title: Institut Paoli Calmettes Hepatic Surgery Database
Acronym: BDD CHIRHEP
Status: Recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: BDD CHIRHEP-IPC 2017-003
Record Dates: First submitted 2018-09-25; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Liver Surgery
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Institut Paoli-Calmettes patients undergoing liver surgery
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Colelction of pre-operative, surgical and post-surgical data

SUMMARY:
Database of patients who undergo hepatic surgery for: benign diseases, primary or secondary liver cancer at Institut Paoli-Calmettes

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing liver surgery for benign liver tumor, primary or secondary liver cancer

Exclusion Criteria:

* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient treated at Institut Paoli-Calmettes who undergo liver surgery for benign liver tumor, primary or secondary liver cancer
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-11-06 (Actual); Primary Completion 2030-11 (Estimated); Study Completion 2030-11 (Estimated)

PRIMARY OUTCOMES:
Epidemiological description | 5 years
  Epidemiological description of the patients who undergo hepatic surgery at Institut Paoli-Calmettes

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Marchese, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches Du Rhone, France

IPD SHARING:
Plan to Share IPD: No